CLINICAL TRIAL: NCT00170755
Title: A Long-Term Safety, Tolerability and Efficacy Study of Darifenacin in Adult Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDAR328A2301
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder, incontinence, antimuscarinic, darifenacin, long-term treatment
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

ARMS (1):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin

INTERVENTIONS:
Drug: Darifenacin — Darifenacin 7,5 mg tablets, Darifenacin 15 mg tablets administered once daily
  Other Names: Enablex

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of darifenacin, in the long-term treatment of adult patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with overactive bladder who completed a previous darifenacin short-term trial.
* Patients capable of independent toileting and able of independently completing the patient diary.

Exclusion Criteria:

* Patients in whom the use of anticholinergic drugs was contraindicated
* Evidence of severe liver disease
* Patients with other clinically significant urinary or gynecological conditions

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2002-04; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Long term safety and tolerability. Safety assessments consisted of monitoring and recording all adverse events (AEs), serious adverse events (SAEs), hematology, blood chemistry, and urinalysis, vital signs, physical condition and body weight.

SECONDARY OUTCOMES:
Long term efficacy on the symptoms of overactive bladder
King's Health questionnaire and EQ-D(at month 3, 6, 12, 24), Patient satisfaction questionnaire, patient valuation questionnaire,bowel questionnaire (at month 6, 12 and 24) and patients' willingness to reuse(at month 12, 24),

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Dwyer P, Kelleher C, Young J, Haab F, Lheritier K, Ariely R, Ebinger U. Long-term benefits of darifenacin treatment for patient quality of life: results from a 2-year extension study. Neurourol Urodyn. 2008;27(6):540-7. doi: 10.1002/nau.20620. PMID 18663723